CLINICAL TRIAL: NCT07017686
Title: The Reboot Study: A Single Group, Open Label Safety Study of Abdominal Vagus Nerve Stimulation for Moderate to Severe Drug Refractory Rheumatoid Arthritis
Brief Title: The Reboot Study: A Safety Study of Abdominal Vagus Nerve Stimulation for Moderate to Severe Drug Refractory Rheumatoid Arthritis
Acronym: Reboot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Bionics Institute of Australia (Other)
Collaborators: St Vincent's Hospital Melbourne (Other); Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 107360; 122/24 (Other: St Vincent's Hospital Melbourne Human Research Ethics Committee)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Arthritis, Rheumatoid
Keywords: Neuromodulation; Inflammatory disease
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: All participants will receive abdominal vagus nerve stimulation (aVNS), delivered by an implanted medical device consisting of an electrode array attached to the abdominal vagus nerve and implantable battery placed under the skin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- abdominal vagus nerve stimulation (aVNS) (Experimental): Participants will receive aVNS, delivered by the implanted aVNS device.
  Interventions: Device: abdominal vagus nerve stimulation (aVNS)

INTERVENTIONS:
Device: abdominal vagus nerve stimulation (aVNS) — Participants will receive aVNS, delivered by a commercially available stimulator placed under the skin, and a custom-designed electrode array attached to the abdominal vagus nerve. Stimulation will commence 2 weeks after laparoscopic surgical implantation of the device, and occur daily for 22-weeks stimulation in the initial phase of the study.
  Other Names: IBDStim; Vagus Nerve Stimulator

SUMMARY:
This open label clinical trial aims to assess the safety of abdominal vagus nerve stimulation (aVNS) for moderate to severe, adult-onset rheumatoid arthritis (RA) that has not responded to medication. The aVNS is an active medical device placed into the body to allow electrical stimulation of the abdominal vagus nerve. Participants will undergo stimulation treatment with the aVNS device from two to 24 weeks after the device is implanted by keyhole surgery. Safety, device performance and potential benefits will be assessed. Participants will be monitored for specific events for 5 years post surgery.

DETAILED DESCRIPTION:
This open label first-in-indication study will assess safety of an abdominal vagus nerve stimulation (aVNS) device in 5 adult participants with moderate to severe drug refractory rheumatoid arthritis (RA). The trial primary objectives at 24 weeks are to assess: 1) safety of aVNS and; 2) device performance. An exploratory objective is to assess non-futile benefits of aVNS at 12 and 24 weeks. During the initial phase of the study (2-24 weeks), stimulation will be delivered for 3 hours per day, with the participant switching the device on and off via a controller. Reports of safety, device checks and clinical assessment of RA symptoms will occur during at 2-, 6-, 12- and 24-weeks post-surgery. Participants that complete the initial phase of the study (24 week assessment) will have the option to continue using the device. Participants that do not want to continue treatment, or withdraw, will have their device deactivated. The device will remain implanted unless there is a clinical reason to remove it or if the participant requests removal. During the follow up phase of the safety trial (24-265 weeks), participants will be monitored twice a year for up to 5 years. The total duration of involvement of participants will be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (18 - 75 years of age).
2. Adult-onset rheumatoid arthritis (RA) (onset age 18 years or above) as defined by the 2010 ACR/EULAR classification criteria, and Rheumatoid Factor (RF) or Cyclic Citrullinated Peptide (CCP) Antibody/Anti-Citrullinated Peptide Antibody (ACPA) must be positive (above lab ranges).
3. Moderate-severe active RA defined by at least 4/28 tender and 4/28 swollen joints.
4. Have active disease that has not responded to a 3-month trial of, or has intolerance limiting a full 3 month trial of, at least 2 biologic and/or new targeted synthetic DMARDs (e.g. JAK inhibitors).
5. Using a stable, continuous dose of at least 1 biological and/or synthetic DMARD for >8 weeks prior to study screening and for the duration of the trial.
6. Women of childbearing age must not be pregnant or trying to become pregnant and must agree to use an effective method of contraception for the duration of their participation in the trial.
7. Medicare eligibility.
8. Provision of informed consent, in the form of a signed and dated informed consent form.

Exclusion Criteria:

1. Unable or unwilling to provide written informed consent.
2. Current diagnosis of major psychiatric disorder/s, or meets criteria as such on the Mini International Neuropsychiatric Interview (MINI), with the exception of stable, well controlled Major Depression or Anxiety Disorder.
3. A medical condition that could interfere with study procedures, and/or confound evaluation of study endpoints, as determined by the Investigator.
4. Medical conditions that have resulted in severe autonomic neuropathy e.g. poorly controlled type 2 diabetes or metabolic disease.
5. History of previous surgical interventions including vagotomy, splenectomy, bariatric surgery.
6. History of gastric hiatus hernia.
7. Previously implanted active medical devices (e.g., dorsal root ganglion or spinal cord stimulators, cardiac pacemakers, automatic implantable cardioverter-defibrillators, drug pumps), or likely need for implantation of such devices within 6 months after start of this study.
8. A condition that requires routine Magnetic Resonance Imaging (MRI) scans
9. Is, in the opinion of the Principal Investigator/s not a suitable candidate for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Safety of aVNS in individuals with drug refractory moderate-severe adult-onset RA. | 24 weeks
  Rate of recorded Serious Adverse Device Effects (SADEs) less than that for the Evoke® device (2%), a commercially available, FDA approved, CE marked implantable spinal cord stimulator.
Safety of aVNS in individuals with drug refractory moderate-severe adult-onset RA. | 24 weeks
  No significant increase in electrically Evoked Compound Action Potentials (ECAPs) threshold
Safety of aVNS in individuals with drug refractory moderate-severe adult-onset RA. | 24 weeks
  No significant decrease in amplitude of electrically Evoked Compound Action Potentials (ECAPs)

SECONDARY OUTCOMES:
Performance of the aVNS System. | 24 weeks
  Rate of device deficiencies less than that for the Evoke® device

OTHER OUTCOMES:
Exploratory Outcome: Non-futile benefits of aVNS in individuals with drug refractory moderate-severe adult-onset RA. | Baseline to week 6, 12 or 24 assessment.
  ACR 20, 50 or 70 response rates in DAS28-CRP from pre-surgery baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Shereen Oon, Principal Investigator — St Vincent's Hospital Melbourne
Locations (3):
- Australia (3):
  - Bionics Institute, Fitzroy, Victoria
  - St Vincent's Hospital, Department of Rheumatology, Fitzroy, Victoria
  - Austin Health, Heidelberg Repatriation Hospital, Ivanhoe, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Payne, S. C., Burns, O., Stebbing, M., Thomas, R., Silva, A. de, Sedo, A., … Shepherd, R. K. (2018). Vagus Nerve Stimulation to Treat Inflammatory Bowel Disease: A Chronic, Preclinical Safety Study in Sheep. Bioelectronics in Medicine, 1(4), 235-250. https://doi.org/10.2217/bem-2018-0011
- [Background] Payne SC, Furness JB, Stebbing MJ. Bioelectric neuromodulation for gastrointestinal disorders: effectiveness and mechanisms. Nat Rev Gastroenterol Hepatol. 2019 Feb;16(2):89-105. doi: 10.1038/s41575-018-0078-6. PMID 30390018
- [Background] Payne SC, Furness JB, Burns O, Sedo A, Hyakumura T, Shepherd RK, Fallon JB. Anti-inflammatory Effects of Abdominal Vagus Nerve Stimulation on Experimental Intestinal Inflammation. Front Neurosci. 2019 May 8;13:418. doi: 10.3389/fnins.2019.00418. eCollection 2019. PMID 31133776
- [Background] Payne SC, Romas E, Hyakumura T, Muntz F, Fallon JB. Abdominal vagus nerve stimulation alleviates collagen-induced arthritis in rats. Front Neurosci. 2022 Nov 21;16:1012133. doi: 10.3389/fnins.2022.1012133. eCollection 2022. PMID 36478876